CLINICAL TRIAL: NCT01023204
Title: Phase II Study of Weekly Paclitaxel (BMS-181339) in Patient With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA139-371
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2009-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; BMS 181339

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel (Experimental)
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — Solution, IV, 100 mg/m², weekly for 6 of 7 weeks, until disease progression or unacceptable toxicity became apparent
  Other Names: Taxol; BMS-181339

SUMMARY:
The purpose of this study is to evaluate the efficacy and the safety of paclitaxel given weekly in patients with advanced or recurrent breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary advanced inoperable disease who were refractory to chemotherapy
* Patients with recurrent disease following post-operative adjuvant chemotherapy
* Patients who were not amenable to post-recurrence chemotherapy

Exclusion Criteria:

* Patients with serious, uncontrolled medical illness
* Patients with previous therapy with taxanes

Ages: 20 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2002-10; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Response rate [defined as total number of patients with complete and partial response divided by number of response-evaluable patients] based on predetermined evaluation criteria | Each 49 day course of treatment until withdrawal or unacceptable toxicity
Safety: incidence and severity of adverse events, laboratory test abnormalities | Each 49 day course of treatment until withdrawal or unacceptable toxicity

SECONDARY OUTCOMES:
Duration of response, defined as either Complete or Partial Response, based on Evaluation Criteria on Therapeutic Effects in Patients with Advanced or Recurrent Breast Cancer | Each 49 day course of treatment until withdrawal or unacceptable toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx